CLINICAL TRIAL: NCT06918509
Title: ASSIST Ethiopia: Feasibility Clinical Investigation of Assisted Vaginal Birth With the Odonassist™ Medical Device
Brief Title: ASSIST Ethiopia: Feasibility Clinical Investigation of the Odonassist™ Medical Device
Acronym: ASSISTEthiopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Doctors with Africa - CUAMM (Other)
Collaborators: Centre Hospitalier Universitaire de Besançon (Unknown); St. Luke Catholic Hospital, Wolisso, Ethiopia (Unknown); Fonds d'Innovation pour le Développement (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CUAMM
Record Dates: First submitted 2025-03-17; First posted 2025-04-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-04

CONDITIONS: Instrumental Delivery; Medical Device; Feasibility Study; Acceptability Study; Pregnancy
Keywords: OdonAssistTM; Instrumental delivery; Medical device; Feasibility study; Acceptability study; pregnancy

STUDY DESIGN:
Intervention Model Description: The ASSIST Ethiopia Study is a feasibility study of women who require an assisted vaginal birth (AVB) for a recognized clinical indication in a low-resource setting.
  Early feasibility studies have reported success rates ranging from 50% to 80%. To ensure we obtain 10 quality assessments from both patients and healthcare providers, a sample size of 20 subjects is anticipated. This number accounts for potential data loss due to technical issues, patient dropouts, and variability in responses. The goal of this feasibility study is to obtain meaningful preliminary data of safety, efficacy and acceptability in a low-resourced setting, that are crucial to inform the implementation of the device within the African environment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OdonAssistTM medical device (Experimental): The ASSIST Ethiopia Study is a feasibility study of women who require an assisted vaginal birth (AVB) for a recognized clinical indication. Assistance will be performed using the OdonAssistTM medical device.
  Interventions: Device: OdonAssistTM

INTERVENTIONS:
Device: OdonAssistTM — Innovative medical device for operative vaginal delivery as an alternative to vacuum or forceps

SUMMARY:
The Innovation The OdonAssist™ is a medical device for assisted vaginal delivery (AVD), that is defined by the need of additional procedure to facilitate childbirth in order to reduce foetal-maternal risks. Increasing access to AVD has been identified by the World Health Organization (WHO) as one of the priorities for improving maternal health globally. The OdonAssist™ is a frugal innovation born in the southern hemisphere in an unconventional environment. It was invented by an Argentinian mechanic, Jorge Odon. Its potential to improve maternal and neonatal health is now recognised. It has been designed to be safe, simple to use and better accepted than current devices (forceps, suction cup). Two studies conducted in England and one in France have confirmed these characteristics and funding has recently been obtained for a randomised clinical investigation in five French hospitals.

Project Rationale The present project aims to conduct a feasibility study at Saint Luke's Hospital in Wolisso, a poorly resourced hospital in rural Ethiopia, in order to test the device in a low-income country and assess its acceptability. In addition, with the aim of investigating the efficiency and budgetary impact of this new device, and considering the wider perspective of a future scale-up, data will be collected on its cost-effectiveness, in order to compare it with the reference interventions at local level (vacuum and caesarean section).

Main research questions:

1. Is it feasible to introduce the OdonAssist™ (new intervention) at the hospital Saint Luke's in Ethiopia, in terms of preliminary data on safety, efficacy, acceptability by mothers and healthcare providers?
2. What are the estimated healthcare-related costs of the OdonAssist™ (new intervention) in comparison to traditional alternatives, that are vacuum-assisted delivery or cesarean section during the second stage of labor?

Study population Participants will be assisted with the OdonAssist™ medical device in case they have provided informed consent and they present medical indication for AVD as per protocol. The study will also collect data on a nested cohort of women and babies delivered either by vacuum extractor or by second-stage cesarean section. The information gained from this study will be used to plan for future impact evaluation and cost utility studies relevant for the implementation and for the scaling up of the OdonAssist™ in low resource settings.

The study site will be Saint Luke's Hospital, Wolisso, Oromia region, Ethiopia.

DETAILED DESCRIPTION:
INTRODUCTION

The OdonAssist™ inflatable device for assisted vaginal birth (AVB), is a frugal innovation from the southern hemisphere and an unconventional environment as it was invented by an Argentinian car mechanic, Jorge Odon. The device has been developed with the intention to be safe, easy to use and more acceptable than currently used AVB devices (forceps and vacuum extractor) because of its innovative mechanism of action. Its potential for improving maternal and neonatal health is now recognized based on the results of three clinical trials conducted in France and UK.

The investigation proposal is to conduct a feasibility study of OdonAssistTM at Saint Luke's Hospital in Wolisso, Ethiopia, to determine the feasibility of using the OdonAssistTM in a low-income country and assess its acceptability in those settings. In addition, with a view to researching the efficiency and budgetary impact of this innovation, data will be collected on its cost and effectiveness, for comparison with reference interventions at local level (vacuum extractor and emergency second stage caesarean section).

Improving the health of mothers and newborns is among the main priorities of the Ethiopian Health Sector Strategic Plan (HSDP IV). The 2016 Ethiopian Demographic and Health Survey preliminary report indicated that Ethiopia has made good progress in reducing neonatal, infant and under five mortalities reporting respectively 29, 48 and 67 deaths per 1,000 live births in years 0-4 prior to the survey, while these figures were 47, 78 and 116 deaths per 1,000 live births 10-14 years prior to the survey. However, the neonatal mortality rate has not declined significantly, nor has the infant and under-five mortality rate and the maternal mortality rate, which is still high at 557 maternal deaths per 100,000 live births caused by pregnancy-related complications (https://data.worldbank.org/indicator/SH.STA.MMRT.NE).

Complications in childbirth are a major cause of maternal and infant mortality and morbidity, accounting for 4-13% of maternal deaths and 25% of neonatal deaths worldwide. Approximately 10-15% of the 134,000,000 births worldwide each year require assistance with forceps or vacuum extractor or emergency caesarean section at full cervical dilation to avoid serious maternal and neonatal complications. In Ethiopia, it is estimated that 12% of pregnant women have a complicated labor, which, according to published studies, causes between 17% and 36% of maternal deaths, 24% of neonatal deaths, 36% of stillbirths and high rates of obstetric fistulas.

The Ethiopian government has made improving maternal and neonatal health a national priority and has identified limited access to AVB as an obstacle to be overcome. The use of innovations has been advocated as a solution to increase access to medical care. These government policies, aimed at improving maternal and newborn health, will be conducive to future efforts to scale up OdonAssistTM in Ethiopia. In addition, the International Federation of Gynecology and Obstetrics (FIGO), which issues globally adopted medical guidelines, has expressed in an official letter its interest in supporting the adoption of OdonAssistTM globally.

PROBLEM STATEMENT AND SIGNIFICANCE OF THE STUDY

Prolonged and complicated labor is a major cause of maternal and neonatal mortality and long-term morbidity. Prolonged or complicated second stage of labor requiring an AVB with forceps or vacuum extractor, or an emergency caesarean section (CS) occurs in approximately 10-15% of births and contributes to 4-13% of all maternal deaths. AVB can be safer than an emergency CS in the short and long term for mothers and babies. AVB is associated with a reduced risk of maternal hemorrhage, intrapartum stillbirth, admission to intensive care for newborns, abnormally invasive placenta (a life-threatening condition for the mother), stillbirth and preterm birth in subsequent pregnancies; AVB is also more cost effective than a cesarean section. The current options for AVB, forceps and vacuum extractor, require time and practice to acquire sufficient skills for use and, if performed inappropriately, can be associated with significant trauma to both mothers and babies. Insufficient training, limited availability of functioning devices, and pervasive concerns about complications are supply side factors that have all reduced access to AVB, particularly in low and middle income countries where there is the most potential benefit (given the growing concentration of maternal & perinatal mortality, as well as the increasing proportion of births, in these settings). Although the World Health OrganisationTM lists AVB as a vital function for all basic emergency obstetric care facilities, African countries commonly report AVB as the least available of these functions. In sub-Saharan African countries, AVB rate is approximately 1% as compared to up to 16% in Western Europe.21 Women living in low resource settings who experience prolonged labor are either: left untreated with dire consequences, or referred for an emergency CS with additional risks associated with the requirement for transfer, the potentially less safe/more invasive surgery and the anesthesia required for laparotomy.29 The OdonAssist™ is an innovation that, because of its innovative simple and potentially less traumatic mechanism of action, is designed to improve women's access to AVB by overcoming the entrenched obstacles and barriers that limit its use with the presently available options of forceps and vacuum extractor.

The mechanism of the OdonAssist is based on inflating an air chamber around the fetal head to act as an anchor point, allowing the practitioner to apply traction. The positive safety profile, as observed in the clinical trials conducted so far, will also reduce the concerns with potential maternal and newborn complications presently associated with AVB. We envisage that, with appropriate but less demanding training than for forceps and vacuum, this device could be used by both doctors and midlevel providers such as midwives when allowed by local laws, health policies and guidelines. In addition, the device is single use and provided sterile and ready to use, thereby eliminating the need to ensure maintenance and functionality.

Given these considerations, the specific aim of the proposed study is to assess the feasibility of the OdonAssist in Ethiopia by collecting preliminary data on efficacy rate, safety profile and acceptability to women and health workers and relate them to the outcomes of AVB with vacuum extractor or cesarean section in the second stage of labor. In addition, data will be collected to inform a future evaluation of the cost utility of the OdonAssist in relation to vacuum and second stage cesarean section.

THE ODONASSIST(TM)

An innovative mechanism of action Because of its innovative mechanism of action, the OdonAssistTM is intended to represent an advance in obstetrics which could enhance the safety of AVB and reduce the training requirements. Differently from the forceps and vacuum extractors, the OdonAssistTM mechanism of action works by inflating an air chamber circumferentially around the fetal head to evenly distribute the pressure needed to establish the anchor point for traction. By using a more flexible and softer anchor point, the pressure is evenly distributed 360 degrees around the fetal head. This mechanism represents a potential advantage relative to the focalized pressure applied by the rigid metal blades of the forceps. The lack of need for negative pressure is expected to reduce the risk of both mild and serious negative-pressure related adverse events associated with vacuum extractors, such as subgaleal hemorrhage. Notably, no typical device related pattern of neonatal superficial injury was observed with the OdonAssist in clinical trials, in contrast to the well-known typical effects seen with the use of forceps (e.g. facial marks) and vacuum extractor (e.g. caput succedaneum and circular bruising). The absence of superficial signs and marks on the baby's head and face associated with the use of AVB devices was appreciated by women and health professionals involved in the clinical studies of OdonAssistTM who reported this differentiating characteristic of OdonAssistTM as one of the reasons to prefer it over forceps.

In addition, the mechanism of action and softness of materials of the OdonAssistTM is likely to cause less pain for the newborn than other AVB devices. Fetal pain receptors and nerve tracts are developed by 20-24 weeks gestation in quantities similar to those found in adults, therefore newborns experience pain which can be assessed using validated pain scales such as the EDIN (Échelle de Douleur Inconfort Nouveau-Née, Neonatal Pain and Discomfort Scale) and the NIPS (Neonatal Infant Pain Scale). AVB with vacuum extractor has been associated with a proportion of EDIN scores indicative of pain (39%) much higher than the levels below 5% reported in the safety and efficacy clinical studies of OdonAssist.

Another important difference and potential advantage of OdonAssist over currently used AVB devices is that the application of OdonAssist is not dependent on the position (occipito-anterior, occipito-transverse and occipito-posterior) of the fetal occiput in the birth canal. The OdonAssist device can be used in all possible occiput positions, therefore increasing ease of use, and minimizing the risk of misapplication. During the clinical trials of the OdonAssist, this characteristic prevented the risk of harming the woman and/or the baby because of incorrect application of the device.

Clinical evidence In the clinical studies conducted until now with the OdonAssistTM, there were no severe adverse events causally related to the device, no serious device-related adverse reactions and no serious adverse device effects. In addition, results emerging from the clinical studies are indicative of high maternal and operator satisfaction and acceptability. Operators found the device easy to use for several reasons including the fact that the same application technique is used for all fetal positions meaning there is no risk of incorrectly positioning the device in relation to vulnerable fetal or maternal anatomies. Satisfaction of mothers regarding the use of the device was very high, as women wanted an alternative device for AVB and were keen for a 'kinder' AVB. The observed effectiveness rate of the device improved progressively over time, increasing in each subsequent study and reaching levels of effectiveness consistent with the range of values for AVB reported in the scientific literature.

STUDY OBJECTIVES

The objectives of the study are:

* To assess the feasibility of the OdonAssist (new intervention) in terms of preliminary data on safety, efficacy, acceptability at the hospital Saint Luke's in Ethiopia and relate them to the performance of vacuum extractor and second stage cesarean section (reference interventions).
* To perform a cost analysis of the OdonAssist (new intervention) at the hospital Saint Luke's in Ethiopia in comparison with vacuum extractor and second stage Cesarean section (reference interventions).

ELIGIBILITY:
Inclusion Criteria:

Women will be able to participate in the ASSIST Ethiopia Study if all of the following apply at initial consent:

* ≥18 years of age;
* singleton pregnancy of at least 36 weeks' gestation,
* negative antenatal screen for HIV and Hepatitis B,
* in active labour and requiring an assisted vaginal birth for a clinical indication (as per local guidelines),
* the vertex is 1 cm or more below the ischial spines and there is no obstetric indication for an alternative method of AVB.

Exclusion Criteria:

Women will not be able to take part in the ASSIST Ethiopia Study if:

* the fetal vertex is at or above the ischial spines,
* there is a diagnosis of a fetal skull abnormality (i.e. macrocephaly) or osteogenesis imperfecta,
* there is a suspicion of a fetal bleeding disorder (von Willebrand's disease, AITP, haemophilia),
* there is an intrauterine fetal death in the current pregnancy,
* the woman is sensitive to latex,
* the woman is currently serving a prison sentence,
* there is a fetal bradycardia which is on-going and has not recovered.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of delivery assistance with the OdonAssistTM medical device | From enrollment to 6 weeks postpartum
  Rate of births successfully assisted with the OdonAssist. An assisted vaginal birth will be defined as 'successful' if all of the following criteria are met:
  * The birth of the baby is expedited with the OdonAssist. (without sequential use of other AVB devices or resorting to cesarean section).
  * There are no serious maternal adverse reactions related to the use of the device during birth.
  * There are no serious neonatal adverse reactions related to the use of the device during birth

SECONDARY OUTCOMES:
Maternal safety - Weighed blood loss (grams) | From enrollment to 6 weeks postpartum
Maternal safety - Perineal and anal sphincter injury | From enrollment to 6 weeks postpartum
  Number of 1st/2nd/3rd/4th degree tears and episiotomy
Maternal safety - Ischio-rectal fossa defect | From enrollment to 6 weeks postpartum
Maternal safety - Cervical tear | From enrollment to 6 weeks postpartum
Maternal safety - cesarean section performed | From enrollment to 6 weeks postpartum
Maternal safety - Maternal death | From enrollment to 6 weeks postpartum
Neonatal safety - Apgar scores at 1, 5 and 10 minutes after birth. | From enrollment to 6 weeks postpartum
  The Apgar scale is a quick assessment of a newborn's well-being after birth, evaluating Appearance (color), Pulse (heart rate), Grimace (reflex irritability), Activity (muscle tone), and Respiration (breathing). Each category is scored 0-2, so total score from 0 to 10 with a higher total score indicating better condition.
Neonatal safety - Shoulder dystocia | From enrollment to 6 weeks postpartum
Neonatal safety - Admission to Neonatal Intensive Care Unit (NICU). | From enrollment to 6 weeks postpartum
Neonatal safety - Duration of admission in NICU (hours). | From enrollment to 6 weeks postpartum
Neonatal safety - Neonatal death | From enrollment to 6 weeks postpartum
Neonatal safety - Neonatal Infant Pain Scores at 2 and 6 h post birth. | From enrollment to 6 weeks postpartum
  Behavioral scale that uses the behaviors that nurses have described as being indicative of infant pain or distress. It is composed of six (6) indicators.
  * facial expression
  * cry
  * breathing patterns
  * arms
  * legs
  * state of arousal Each indicator is scored with 0 or 1 except "cry", which has three possible descriptors therefore, being scored with a 0, 1 or 2. See the NIPS scale for the description of infant behavior in each indicator group. Infants should be observed for one minute in order to fully assess each indicator. Total pain scores range from 0-7. The suggested interventions based upon the infant's level of pain are listed below.
  0-2 = mild to no pain - No intervention 3-4 = mild to moderate pain - Non-pharmacological intervention, reassessment in 30 minutes >4 = severe pain - Non-pharmacological intervention and possibly a pharmacological intervention with reassessment in 30 minutes
Neonatal safety - Neonatal soft tissue trauma | From enrollment to 6 weeks postpartum
  bruise/scalp injury/facial injury/cephalohaematoma
Neonatal safety - other neonatal complication | From enrollment to 6 weeks postpartum
  subaponeurotic haemorrhage/hematoma/bone fracture/cerebral contusion/neurological sign/seizure/phototherapy for jaundice/organ failure
Birth related outcomes - Time from 'decision to perform assisted birth' to 'birth' (minutes). | From enrollment to 6 weeks postpartum
Birth related outcomes - Time from 'device application" to 'birth' (minutes). | From enrollment to 6 weeks postpartum
Birth related outcomes - Location of birth. | From enrollment to 6 weeks postpartum
  operating room/delivery ward
Birth related outcomes - Mode of birth following failed use of OdonAssist. | From enrollment to 6 weeks postpartum
  vacuum assisted/forceps assisted/second-stage cesarean section
Device-related outcomes - Failure of a component of the OdonAssist. | From enrollment to 6 weeks postpartum
  number, description of component the failure was attributed to
Device-related outcomes - Number of applications of device. | From enrollment to 6 weeks postpartum
Device-related outcomes - Number of pulls of the device. | From enrollment to 6 weeks postpartum
Device-related outcomes - Perceived reason for device failure from operator | From enrollment to 6 weeks postpartum
  descriptive, can be attributed to maternal/clinical/device/other factor
Patient-reported outcomes - Maternal health-related quality of life data (EQ-5D-5L) at day 1 postnatal. | From enrollment to 6 weeks postpartum
  The Maternal health-related quality of life (HRQoL) data using the EQ-5D-5L scale is a brief, standardized questionnaire assessing five dimensions of health (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each with five levels of severity (from 0 to 4, from worse to good health). The overall health state can be converted to a single index score, with the range being 0 to 20, where 20 represents full health and 0 value indicate health states considered worse than death. Additionally, a visual analogue scale (VAS) from 0 (worst imaginable health) to 100 (best imaginable health) is included for a direct self-rating of current health.
Patient-reported outcomes - Maternal perception of pain at day 1 postnatal | From enrollment to 6 weeks postpartum
  Perception of pain on an 11-point Likert scale is a subjective self-report where individuals rate their pain intensity on a numerical range from 0 (no pain) to 10 (worst imaginable pain).
Acceptability of the OdonAssistTM medical device - Woman acceptability will be assessed through the patient perception score of birth experience on days 1 postnatal and through qualitative assessment | From enrollment to 6 weeks postpartum
  Patient's perception of birth experience: score out of 15 where 3 is the lowest score possible and 15 maximum.
  * I felt safe during birth (from 1 to 5, 1 worst and 5 best subjective experience)
  * I felt informed during birth (from 1 to 5, 1 worst and 5 best subjective experience)
  * I felt respected during birth (from 1 to 5, 1 worst and 5 best subjective experience) The patient will also be interviewed to collect descriptive information about birth experience
Acceptability of the OdonAssistTM medical device - Practitioner acceptability will be assessed through perceived outcomes following each attempted AVB. | From enrollment to 6 weeks postpartum
  The following will be collected on a 5-point Likert scale (from 1 to 5, worst to best experience) :
  * Perceived overall ease of use of device (for all AVBs).
  * Ease of device set-up (for all AVBs).
  * Ease of device application to the baby's head (for all AVBs).
  * Ease of withdrawal of the applicator after application (for OdonAssist).
  * Comfort with the level of force required to assist the birth of thebaby (for all AVBs).
  * Ease of deflation of the cuff prior to crowning (for OdonAssist).
  * Ease of removal of vacuum extractor. Total score from 7 to 35, worst to best experience.
Health economics - Health care resource use and associated health care costs (USD) | From enrollment to 6 weeks postpartum
  * Direct medical costs will included costs related to treatment (hospitalization, in- and out-patient treatments), monitoring (clinical, biological), medical consultations and management of complications.
  * Indirect medical and intangible costs will be not analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Bobbio, MD, Principal Investigator — Doctors with Africa - CUAMM
Locations (1):
- St. Luke Catholic Hospital, Waliso, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
The opportunity to share individual participant data will be discussed with all relevant partners involved in the study.

REFERENCES:
- [Background] Schuller C, Kanel N, Muller O, Kind AB, Tinner EM, Hosli I, Zimmermann R, Surbek D. Stress and pain response of neonates after spontaneous birth and vacuum-assisted and cesarean delivery. Am J Obstet Gynecol. 2012 Nov;207(5):416.e1-6. doi: 10.1016/j.ajog.2012.08.024. Epub 2012 Aug 17. PMID 22959831
- [Background] Hotton EJ, Blencowe NS, Lenguerrand E, Draycott TJ, Crofts JF, Wade J. Women's experiences of the Odon Device to assist vaginal birth and participation in intrapartum research: a qualitative study in a maternity unit in the Southwest of England. BMJ Open. 2021 Dec 15;11(12):e057023. doi: 10.1136/bmjopen-2021-057023. PMID 34911726
- [Background] Sobhy S, Arroyo-Manzano D, Murugesu N, Karthikeyan G, Kumar V, Kaur I, Fernandez E, Gundabattula SR, Betran AP, Khan K, Zamora J, Thangaratinam S. Maternal and perinatal mortality and complications associated with caesarean section in low-income and middle-income countries: a systematic review and meta-analysis. Lancet. 2019 May 11;393(10184):1973-1982. doi: 10.1016/S0140-6736(18)32386-9. Epub 2019 Mar 28. PMID 30929893
- [Background] Verma GL, Spalding JJ, Wilkinson MD, Hofmeyr GJ, Vannevel V, O'Mahony F. Instruments for assisted vaginal birth. Cochrane Database Syst Rev. 2021 Sep 24;9(9):CD005455. doi: 10.1002/14651858.CD005455.pub3. PMID 34559884
- [Background] Bahl R, Hotton E, Crofts J, Draycott T. Assisted vaginal birth in 21st century: current practice and new innovations. Am J Obstet Gynecol. 2024 Mar;230(3S):S917-S931. doi: 10.1016/j.ajog.2022.12.305. Epub 2023 Jul 28. PMID 38462263
- [Background] Moraitis AA, Oliver-Williams C, Wood AM, Fleming M, Pell JP, Smith G. Previous caesarean delivery and the risk of unexplained stillbirth: retrospective cohort study and meta-analysis. BJOG. 2015 Oct;122(11):1467-74. doi: 10.1111/1471-0528.13461. Epub 2015 May 29. PMID 26033155
- [Background] Clark EA, Silver RM. Long-term maternal morbidity associated with repeat cesarean delivery. Am J Obstet Gynecol. 2011 Dec;205(6 Suppl):S2-10. doi: 10.1016/j.ajog.2011.09.028. Epub 2011 Oct 6. PMID 22114995
- [Background] Bailey PE, van Roosmalen J, Mola G, Evans C, de Bernis L, Dao B. Assisted vaginal delivery in low and middle income countries: an overview. BJOG. 2017 Aug;124(9):1335-1344. doi: 10.1111/1471-0528.14477. Epub 2017 Jan 31. PMID 28139878
- [Background] Nolens B, Capelle M, van Roosmalen J, Mola G, Byamugisha J, Lule J, Faye A, van den Akker T. Use of assisted vaginal birth to reduce unnecessary caesarean sections and improve maternal and perinatal outcomes. Lancet Glob Health. 2019 Apr;7(4):e408-e409. doi: 10.1016/S2214-109X(19)30043-9. No abstract available. PMID 30879501
- [Background] Maheu-Giroux M, Filippi V, Samadoulougou S, Castro MC, Maulet N, Meda N, Kirakoya-Samadoulougou F. Prevalence of symptoms of vaginal fistula in 19 sub-Saharan Africa countries: a meta-analysis of national household survey data. Lancet Glob Health. 2015 May;3(5):e271-8. doi: 10.1016/S2214-109X(14)70348-1. PMID 25889469
- [Background] Gedefaw G, Wondmieneh A, Getie A, Bimerew M, Demis A. Estimating the Prevalence and Risk Factors of Obstetric Fistula in Ethiopia: Results from Demographic and Health Survey. Int J Womens Health. 2021 Jul 7;13:683-690. doi: 10.2147/IJWH.S306221. eCollection 2021. PMID 34262358
- [Background] Berhan Y, Berhan A. Causes of maternal mortality in Ethiopia: a significant decline in abortion related death. Ethiop J Health Sci. 2014 Sep;24 Suppl(0 Suppl):15-28. doi: 10.4314/ejhs.v24i0.3s. PMID 25489180
- [Background] Ayenew AA. Incidence, causes, and maternofetal outcomes of obstructed labor in Ethiopia: systematic review and meta-analysis. Reprod Health. 2021 Mar 10;18(1):61. doi: 10.1186/s12978-021-01103-0. PMID 33691736
- [Background] Addisu D, Mekie M, Melkie A, Yeshambel A. Burden of obstructed labor in ethiopia: A systematic review and meta-analysis. Midwifery. 2021 Apr;95:102930. doi: 10.1016/j.midw.2021.102930. Epub 2021 Feb 5. PMID 33581417
- [Background] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Background] Mottet N, Hotton E, Eckman-Lacroix A, Bourtembourg A, Metz JP, Cot S, Poitrey E, Delhomme L, Languerrand E, Nallet C, Lallemant M, Draycott T, Riethmuller D. Safety and efficacy of the OdonAssist inflatable device for assisted vaginal birth: the BESANCON ASSIST study. Am J Obstet Gynecol. 2024 Mar;230(3S):S947-S958. doi: 10.1016/j.ajog.2023.05.016. Epub 2023 Aug 1. PMID 38462265
- [Background] Hotton EJ, Bale N, Rose C, White P, Wade J, Mottet N, Loose AJ, Elhodaiby M, Lenguerrand E, Draycott TJ, Crofts JF; ASSIST II Study Group. The OdonAssist inflatable device for assisted vaginal birth-the ASSIST II study (United Kingdom). Am J Obstet Gynecol. 2024 Mar;230(3S):S932-S946.e3. doi: 10.1016/j.ajog.2023.05.018. Epub 2023 Jul 30. PMID 38462264
- [Background] Hotton EJ, Lenguerrand E, Alvarez M, O'Brien S, Draycott TJ, Crofts JF; ASSIST Study Team. Outcomes of the novel Odon Device in indicated operative vaginal birth. Am J Obstet Gynecol. 2021 Jun;224(6):607.e1-607.e17. doi: 10.1016/j.ajog.2020.12.017. Epub 2020 Dec 13. PMID 33316274